CLINICAL TRIAL: NCT04315844
Title: The Trial of Ewata Balloon Guiding in the Application of Thrombectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Zhongrong Miao, Chief physician, Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCXY-02-01
Record Dates: First submitted 2020-03-18; First posted 2020-03-20 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Acute Ischemic Stroke
Keywords: AIS balloon guiding
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- balloon (Experimental): To evaluate the efficacy and security of Ewata combined with a stent device in the treatment of acute ischemic stroke within 8 hours To prove whether the clinical efficacy and safety of Ewata r is not inferior to other guidings.
  Interventions: Device: Ewata balloon guiding

INTERVENTIONS:
Device: Ewata balloon guiding — The balloon guide catheter is coaxial cavity and reinforced braided catheter with varying stiffness echelon.The distal end is marked by an impermeable ray, the proximal end has a bifurcated ruhr interface, and the end is embedded with a compliance balloon.The product label indicates the size of the balloon guide catheter and the maximum volume of the balloon.

SUMMARY:
To evaluate the efficacy and security of Ewata combined with a stent device in the treatment of acute ischemic stroke within 8 hours To prove whether the clinical efficacy and safety of Ewata r is not inferior to other guidings.

DETAILED DESCRIPTION:
This clinical trial uses multicenter, single-arm, prospective trial design,people who met the enrollment requirements were performed with Ewata balloon guiding and stent type thrombectomy device.The clinical results were compared with those of other historical guiding catheter products combined with the stent type thrombectomy device to to evaluate the clinical efficacy and safety of Ewata balloon guide catheter in combination with a stent for thrombectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke
2. within 8 hours
3. Patients aged 18-80 years (including critical point)
4. NIHSS score 4-30 (including critical points)
5. Pre-onset mRS score <2
6. Large vessel lesions were detected by head CT, CTA, MRI, MRA, or DSA
7. The patient or his legal guardian voluntarily signs and dates a written informed 8.consent approved by the ethics committee (IBC).

Exclusion Criteria:

1. Head CT exclusion criteria (exclusion if any of the following conditions are met)
2. Cerebral hemorrhage
3. Intracranial tumors, except for small meningiomas
4. Large area of early cerebral infarction (low density shadow >1/3 cerebral hemisphere)

Clinical and laboratory exclusion criteria

1. seizure
2. Symptoms of nervous system loss improved rapidly
3. Severe stroke (NIHSS≥31 points) or mild stroke (NIHSS≤3 points)
4. CT examination of the skull was negative, but subarachnoid hemorrhage was not excluded from clinical symptoms
5. A history of intracranial hemorrhage and subarachnoid hemorrhage
6. A history of cranial trauma in the last 3 months
7. A history of cerebral or myocardial infarction in the last 3 months
8. A history of gastrointestinal or urinary tract bleeding in the last 3 weeks
9. A history of major surgery in the last 2 weeks
10. A history of arterial puncture in the last l weeks that was difficult to stop bleeding
11. Patients with severe cardiac, hepatic or renal insufficiency (>250 mol/L) or severe diabetes mellitus
12. Physical examination revealed evidence of active bleeding or trauma, such as a fracture
13. Oral anticoagulants have been taken, and INR>1.7
14. Blood glucose <2.7 mmol/L or >22.2 mmol/L
15. Systolic blood pressure >185 mmHg, or diastolic blood pressure >110 mmHg Pregnancy
16. There is a tendency of severe bleeding or bleeding disease, platelet count ≤80x109 /L
17. Systemic infection without control or local infection of puncture point Hypersensitivity to contrast media

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
technical success rate of ewata | intraoperative
  When the balloon guiding catheter arrives at the desired location, the thrombectomy instrument can enter the balloon guiding catheter smoothly, which can be opened successfully when needed to form a local blockage of blood flow. After the thrombectomy, the thrombectomy instrument can be withdrawn back into the guide catheter, which is considered as a success.Ewata balloon guide catheter should be used at least once during thrombectomy

SECONDARY OUTCOMES:
Rate of Vascular recanalization | postoperative
  TICI≥2b
Rate of intraoperative adverse events | intraoperative
  including vascular perforation , incision,vasospasm caused by balloon guiding,balloon guide catheter rupture and other instrument-related accidents
The time from the successful puncture to the expected location of ewata | intraoperative
  time data
The time from successful puncture to recanalization | intraoperative
  time data,TICI≥2b
Rate of symptomatic intracranial hemorrhage within 24 hours | 24 hours
  CT/NIHSS
24-hour mortality | 24-hour
  The number of all deaths reported will be recorded and adjudicated
90-day mortality | 90-day
  The number of all deaths reported will be recorded and adjudicated
Good prognosis rate at 90 days | 90 days
  (mRS≤2)
The thrombus escapes from the target vessel to other vessels to form new embolism | intraoperative
  The form of New thrombosis Judged by DSA or MRA

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China